CLINICAL TRIAL: NCT00662987
Title: Effect of Duration of Antibiotic Therapy on Recovery Following Tonsillectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Jacqueline Jones, MD, Department of Otorhinolaryngology, Weill Cornell Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WCMC0506007924
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2008-04-21 (Estimated); Status verified 2008-04

CONDITIONS: Tonsillectomy
Keywords: tonsillectomy; antibiotics
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group B (Placebo Comparator): Received 3 days of amoxicillin followed by 4 days of placebo
  Interventions: Drug: 3 days of amoxcillin followed by 4 days of placebo
- Group A (Active Comparator): Received 7 days of amoxicillin
  Interventions: Drug: 7 days of amoxicillin

INTERVENTIONS:
Drug: 7 days of amoxicillin — Received 7 days of amoxicillin (dosed 40mg/kg divided bid up to maximum daily dose of 800 mg)
  Arms: Group A
Drug: 3 days of amoxcillin followed by 4 days of placebo — 3 days of amoxicillin (40 mg/kg divided bid up to maximum daily dose of 800 mg) followed by placebo
  Arms: Group B

SUMMARY:
To determine whether a 3-day course of postoperative antibiotics is effective as a 7-day course in reducing pain and reducing time to resumption of normal diet and activity following pediatric tonsillectomy

DETAILED DESCRIPTION:
STUDY DESIGN : A prospective, randomized, placebo-controlled trial METHODS : All pediatric patients (under the age of 18) scheduled to undergo a tonsillectomy with or without adenoidectomy from an outpatient otolaryngology practice will be recruited for the study. Exclusion criteria include prior use of antibiotics 7 days before surgery, penicillin allergy or medical comorbidity necessitating antibiotic use. Preoperative demographic information will be obtained. Tonsillectomy with or without adenoidectomy will be performed by a single surgeon (JJ) using electrocautery. Patients will be randomized to receive either a 3- or 7-day course of amoxicillin. Parents will be asked to record the following information: analgesic use for the first 7 postoperative days, postoperative days the child initiated her usual diet and level of activity and medical treatment for oral hemorrhage or dehydration. Statistical analysis will be performed to determine a real difference between the two groups with regard to analgesic use, resumption to normal diet and activity, and incidence of oral hemorrhage or dehydration.

ELIGIBILITY:
Inclusion Criteria:

* tonsillectomy with or without adenoidectomy
* under the age of 18

Exclusion Criteria:

* penicillin allergy
* took antibiotics within 7 days of surgery
* medical comorbidity requiring treatment with antibiotics

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2005-09; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
analgesic use | 1 week

SECONDARY OUTCOMES:
time of resumption of normal diet | 1 week
time of resumption of normal activity | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Jones, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Derived] Johnson PE, Rickert SM, Jones J. Duration-related efficacy of postoperative antibiotics following pediatric tonsillectomy: a prospective, randomized, placebo-controlled trial. Arch Otolaryngol Head Neck Surg. 2009 Oct;135(10):984-7. doi: 10.1001/archoto.2009.146. PMID 19841335